CLINICAL TRIAL: NCT07372846
Title: Evaluation of the Correlation Between Body Roundness Index (BRI), Body Mass Index (BMI), and VIDAC Score in Obese Patients: A Prospective Observational Study
Brief Title: BRI, BMI, and VIDAC Score Relationship in Obese Patients
Acronym: BRI-VIDAC
Status: Recruiting | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: GOKAEK 2025/23/18
Record Dates: First submitted 2026-01-02; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Vidiac Score
Keywords: obesity; vidiac score; videolaryngoscopy; body mass index; Body Roundness Index
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: Correlation between videolaryngoscopy imaging score and body mass index.
  Interventions: Device: VIDEOLARYNGOSCOPE
- group 2: Correlation between videolaryngoscopy imaging score and body roundness index .
  Interventions: Device: VIDEOLARYNGOSCOPE

INTERVENTIONS:
Device: VIDEOLARYNGOSCOPE — Videolaryngoscopy imaging in participants with a body mass index greater than 30 kg/m².

SUMMARY:
The VIDIAC score is a measurement system that objectively defines glottic visibility and anatomical complexity in videolaryngoscopy. The literature has shown a relationship between parameters such as BMI, NC, and TMD and difficult airway management in obese patients, but there is no study examining the BRI-VIDIAC relationship.

DETAILED DESCRIPTION:
Obesity is a clinical condition that alters the anatomical airway structure and can increase intubation difficulties.

Body Mass Index (BMI) alone is not a sufficient predictor of airway management; it is important in conjunction with measurements such as obesity-related fat distribution, neck circumference, and temporomandibular joint dysfunction (TMD). Body Roundness Index (BRI) is a new anthropometric indicator that reflects body fat distribution more accurately than BMI.

The VIDIAC score is a measurement system that objectively defines glottic visibility and anatomical complexity in videolaryngoscopy. The literature has shown a relationship between parameters such as BMI, NC, and TMD and difficult airway management in obese patients, but there is no study examining the BRI-VIDIAC relationship.

This study aimed to examine the correlation of BRI and BMI values with the VIDIAC score and to determine whether BRI is a stronger predictor of difficult airway management than BMI.

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia will be administered
* Being classified as obese (BMI ≥30)
* Patient giving informed consent

Exclusion Criteria:

* Pregnancy
* Emergency surgery
* Head and neck deformity
* Inability to measure Mallampati level
* Patients with tracheostomy
* Severe hemodynamic instability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged 18-65 with a BMI ≥ 30 kg/m² who will undergo elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Examining the correlation between BRI and BMI values and the VIDIAC score. | 3 minutes after anesthesia induction
  To examine the correlation between BRI and BMI values and the VIDIAC score, and to determine whether BRI is a stronger predictor of difficult airway passage than BMI.

SECONDARY OUTCOMES:
number of intubation attempts | 3 minutes after anesthesia induction
  To evaluate the relationship between BRI and BMI and the number of intubation attempts.
Oropharyngeal visibility | 3 minutes after anesthesia induction
  To examine its relationship with oropharyngeal visibility (Cormack-Lehane, Mallampati).

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun University, Samsun Training and Research Hospital, Samsun, Ilkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request